CLINICAL TRIAL: NCT06229431
Title: Supporting Older Spousal Caregivers Who Care for a Partner With Multimorbidity at Home - a Cluster Randomized Person-centred Intervention Trial to Promote Preparedness, Quality of Life and Health
Brief Title: Supporting Older Spousal Caregivers Who Care for a Partner With Multimorbidity at Home
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Maria Norinder, Project coordinator, Ersta Sköndal University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ErstaSUC3
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Family Members; Home Care Services; Support, Family

STUDY DESIGN:
Intervention Model Description: This intervention study has a cluster-randomised design developed in accordance with the CONSORT statement
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSNAT intervention (Experimental): District nurses will be trained to use the CSNAT-I on family caregivers to persons with multimorbidity at home.
  Interventions: Other: The Carer Support Needs Assessment Tool Intervention (CSNAT-I)
- Control (No Intervention): Standard support and care.

INTERVENTIONS:
Other: The Carer Support Needs Assessment Tool Intervention (CSNAT-I) — The CSNAT tool The tool includes 16 questions about the need for more support.
  The five-stage person-centered approach
  In the present study, the CSNAT-I consist of at least two meetings between the older spousal caregiver and the district nurse,1-4 weeks apart, following 5 stages:
  1. Introduction of the CSNAT tool as a conversation starter.
  2. Time for the spousal caregiver to consider the questions in which more support is needed.
  3. An assessment conversation takes place.
  4. A shared action plan is formed based on the assessment conversation.
  5. Continuous shared review of the action plan.
  Arms: CSNAT intervention

SUMMARY:
Research problem and specific questions:

This project aims to evaluate the person-centred Carer Support Needs Assessment Tool Intervention (C SNAT-I), in Swedish "Ditt behov av stöd". The project goal is to promote preparedness, quality of life and health for older spousal caregivers (≥65 years) who care for a partner (≥65years) with multimorbidity at home.

Data, method and plan for realisation:

With a cluster randomised controlled design in a primary health care context the C SNAT-I will be tested. The intervention consists of two parts, an evidence-based tool and a personcentred five stage process to proactively identify and address caregivers needs: 1) introduction of the CSNAT tool comprising 16 questions about the need for support, 2) caregiver consideration and reflection on support needs, 3) an assessment conversation between the caregiver and a nurse, 4) a shared action plan is formed and 5) continuous review of support needs and action plan. Primary health care centres will be randomized to intervention or control arm. Multiple research methods for data collection and analyses will be used. In total 180 caregivers will be recruited for one year and data collected at baseline, 8 and 16 weeks later.

DETAILED DESCRIPTION:
Research problem and specific questions: This project aims to evaluate the person-centred Carer Support Needs Assessment Tool Intervention (CSNAT-I), in Swedish "Ditt behov av stöd". The project goal is to promote preparedness, quality of life and health for older spousal caregivers (≥65 years) who care for a partner (≥65 years) with multimorbidity at home.

Data, method and plan for realisation: With a cluster randomised controlled design in a primary health care context the CSNAT-I will be tested. The intervention consists of two parts, an evidence-based tool and a person-centred five stage process to proactively identify and address caregivers needs: 1) introduction of the CSNAT tool comprising 16 questions about the need for support, 2) caregiver consideration and reflection on support needs, 3) an assessment conversation between the caregiver and a nurse, 4) a shared action plan is formed and 5) continuous review of support needs and action plan. Primary health care centres will be randomized to intervention or control arm. Multiple research methods for data collection and analyses will be used. In total 180 caregivers will be recruited for one year and data collected at baseline, 8 and 16 weeks later. The realisation of the project is strengthened by previous research and the current collaboration between researchers at four universities, the Academic Primary Health Care Centre, Stockholm Gerontology Research Center, a care consultant and a caregiver representative.

Social relevance and utilisation: National and international studies have shown the CSNAT-I to be beneficial for both family caregivers and health care professionals in specialised home care. The CSNAT tool and a training toolkit for health care professionals including guidance about how to work with the intervention is available in Swedish. The intervention is successfully tested in specialised palliative home care in Sweden. Given older spousal caregivers need of support, it is vital to evaluate the CSNAT-I in the new context of primary home health care. This is important as primary health care is emphasized as the foundation stone in Swedish health care according to the national guidelines of "Nära vård". The project ties in with the first "Nationella anhörigstrategi" which aims at promoting support for family caregivers. If preparedness, quality of life and health is found to be promoted, the CSNAT-I can be used to support older caregivers proactively and systematically.

ELIGIBILITY:
Inclusion Criteria:

Older spousal caregivers, who cares for a partner (≥65 years) diagnosed with multimorbidity and admitted to primary home health care, are to be included in the study. Caregivers should be ≥65 years and understand and speak the Swedish language.

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Preparedness for Caregiving Scale (PCS) | Data will be collected at baseline (before the CSNAT-I) and follow-up, 8 and 16 weeks after completed CSNAT-I.
  The scale will be used to measure changes in caregiver's self-reported predparedness for caregiving. The scale consists of eight items answered on a five-point Likert-type response scale ranging from 'Not at all prepared' (0) to 'Very well prepared' (4). The responses are summed into a total score with a possible range between 0 and 32.

SECONDARY OUTCOMES:
The Quality of Life in Life-Threatening Illness Family caregiver version (QOLLTI-F) | Data will be collected at baseline (before the CSNAT-I) and follow-up, 8 and 16 weeks after completed CSNAT-I.
  The scale will be used to measure changes in caregiver's self-reported quality of life. The scale consists of a total of 17 items divided into 7 subscales assessing different domains of quality of life: Environment, Patient condition, Family caregiver's own state, Family caregiver's outlook, Quality of care, Relationships, and Financial worries. It also includes 1 item about overall Quality of life. All items are scored on an 11-point numeric rating scale, ranging between 0-10 with a descriptive anchor at each extreme. Each domain is calculated by adding the responses and dividing the sum by the number of items in each domain. Thus, each domain can range between 0-10, and after reversed items have been rescored, higher scores indicate higher levels of quality of life
General health subscale from RAND-36 | Data will be collected at baseline (before the CSNAT-I) and follow-up, 8 and 16 weeks after completed CSNAT-I.
  The scale will be used to measure changes in in caregiver's self-reported health. For this study we have choosen to use a single item measuring general health. The item is calculated on a five point scale, ranging from 1-5, where higher values indicate better health.
The Carer Support Needs Assessment Tool (CSNAT) | Data will be collected at baseline (before the CSNAT-I) and follow-up, 8 and 16 weeks after completed CSNAT-I.
  The scale will be used to measure changes in caregiver's self-reported support needs. The instrument consists of 16 domains/questions. The CSNAT has three response categories indicating how much more support caregivers need, ranging from 'no more support' to 'very much more support'. The CSNAT is not developed to be summed into a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Alvariza, PhD, Principal Investigator — Marie Cedershiöld University
Locations (1):
- Marie Cederschiöld University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No